CLINICAL TRIAL: NCT00483015
Title: Differences in the Presentation, Outcome and Response to Treatment Between Never- Smokers and Smokers With Non- Small Cell Lung Cancer.
Brief Title: Differences in the Presentation Outcome and Response to Treatment Between Never- Smokers and Smokers With NSCLC
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 05-0707
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Smokers
Keywords: presentation; outcome; response; never- smokers
MeSH Terms: interventions — Smoking Devices

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: smoking

SUMMARY:
We wish to discover if there is a difference in the presentation, response to treatment and survival of never- smokers with lung cancer as compared to ever- smokers.

We also plan to obtain tumor specimens to compare the genetic and proteomic expression between smokers and never smokers

DETAILED DESCRIPTION:
Lung cancer is the most lethal of all malignant tumors affecting humans. In the United States alone an estimated 160,440 patients died of lung cancer 2004[1]. It is well known that tobacco smoking is a major risk factor and accounts for the majority of all lung cancer cases. But there is a sub group of patients with lung cancer who have never actively smoked tobacco. This group exhibits certain unique characteristics which separates them from lung cancer in smokers. It has been shown that never- smokers with adenocarcinoma have better outcomes in terms of overall survival as well as lung cancer specific survival when compared to current smokers with adenocarcinoma of the lung[2]. Also patients who are current smokers at diagnosis have decreased survival when compared to people who quit smoking[3]. The improved survival in never smokers could be due to several reasons. Such as increased incidence of co-morbid factors in smokers as result of exposure to tobacco smoke, differences in metabolism of chemotherapeutic agents or a reflection of differences in the underlying molecular biology of the tumor.

It has been demonstrated that chromosomal abnormalities are common in lung cancer patients with a smoking history when compared to never- smokers[4]. Gene mutations such as p53 mutations are more frequent in never- smokers than in previous smokers[5]. In addition mutations that are specific only to lung cancer in never smokers have been discovered, demonstrating the possibility of a separate or overlapping carcinogenesis pathway for lung cancer in never smokers vs. smokers [6].

ELIGIBILITY:
Inclusion Criteria:

* Age Range 18-88, diagnosed with non- small cell lung cancer between Jan 1 1996 and Dec 31 2002.

Exclusion Criteria:

* Patients diagnosed prior to Dec 31, 1995 and after Jan 1, 2003

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age Range 18-88, diagnosed with non- small cell lung cancer between Jan 1 1996 and Dec 31 2002.
Enrollment: 280 (Actual)
Dates: Start 2006-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Tammemagi CM, Neslund-Dudas C, Simoff M, Kvale P. Impact of comorbidity on lung cancer survival. Int J Cancer. 2003 Mar 1;103(6):792-802. doi: 10.1002/ijc.10882. PMID 12516101
- [Background] Sanchez-Cespedes M, Ahrendt SA, Piantadosi S, Rosell R, Monzo M, Wu L, Westra WH, Yang SC, Jen J, Sidransky D. Chromosomal alterations in lung adenocarcinoma from smokers and nonsmokers. Cancer Res. 2001 Feb 15;61(4):1309-13. PMID 11245426
- [Background] Vahakangas KH, Bennett WP, Castren K, Welsh JA, Khan MA, Blomeke B, Alavanja MC, Harris CC. p53 and K-ras mutations in lung cancers from former and never-smoking women. Cancer Res. 2001 Jun 1;61(11):4350-6. PMID 11389059
- [Background] Gazdar AF. Lung cancer in never smokers - A different pathway. ASCO 2005:619-21
- [Result] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Result] Nordquist LT, Simon GR, Cantor A, Alberts WM, Bepler G. Improved survival in never-smokers vs current smokers with primary adenocarcinoma of the lung. Chest. 2004 Aug;126(2):347-51. doi: 10.1378/chest.126.2.347. PMID 15302716
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu